CLINICAL TRIAL: NCT06728748
Title: Retrospective Multicentre Study on the Impact of Neonatal Screening for Congenital Adrenal Hyperplasia in Italy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ISCREEN
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Oservational, retrospective, multicenter study focused on neonatal screening for Congenital Adreanl Hyperplasia.

DETAILED DESCRIPTION:
The study refers to neonates who underwent neonatal screening for Congenital Adreanl Hyperplasia between January 2006 and December 2019 at participating centres, but only patients diagnosed with Congenital Adreanl Hyperplasia are enrolled in the study.

The primary aims are: to assess the incidence of classic Congenital Adrenal Hyperplasia in neonates who underwent neonatal screening in the reporting period; to calculate the sensibility of Neonatal Screening for classic Congenital Adrenal Hyperplasia; to calculate the positive predictive rate. The secondary aims are: to describe the biochemical, hormonal, and clinical features of neonates at diagnosis of Congenital Adrenal Hyperplasia; to assess the time required for diagnosis; to calculate the false positive rate; to calculate the diagnostic impact of neonatal screening for Congenital Adrenal Hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal who underwent neonatal screening for congenital adrenal hyperplasia between January 2006 and December 2019 at participating centres;
* Patients diagnosed with Congenital Adrenal Hyperplasia;
* Obtaining informed consent.

Exclusion Criteria:

• None.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study refers to neonates who underwent neonatal screening for Congenital Adreanl Hyperplasia between January 2006 and December 2019 at participating centres, but only patients diagnosed with Congenital Adreanl Hyperplasia are enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of classic Congenital Adrenal Hyperplasia in neonates who underwent neonatal screening in the reporting period | at baseline
  number of patients diagnosed with classic Congenital Adrenal Hyperplasia between January 2006 and December 2019
Sensibility of Neonatal Screening for classic Congenital Adrenal Hyperplasia | at baseline
  Sensibility of Neonatal Screening
Positive predictive rate | at baseline
  TP / (TP + FP)

SECONDARY OUTCOMES:
Neonatal clinical features at diagnosis of Congenital Adrenal Hyperplasia | at baseline
  gestational age (weeks)
Neonatal clinical features at diagnosis of Congenital Adrenal Hyperplasia | at baseline
  neonatal weight (g)
Neonatal biochemical features at diagnosis of Congenital Adrenal Hyperplasia | at baseline
  serum electrolytes
Neonatal hormonal features at diagnosis of Congenital Adrenal Hyperplasia | at baseline
  blood renin value (microU/mL)
Neonatal hormonal features at diagnosis of Congenital Adrenal Hyperplasia | at baseline
  blood plasma values of 17α-hydroxyprogesterone (ng/dL)
Time required for diagnosis of Congenital Adrenal Hyperplasia | at baseline
  Time required for diagnosis
False positive rate | at baseline
  TP / (TP + FP)
Diagnostic impact of neonatal screening for Congenital Adrenal Hyperplasia | at baseline
  ratio between the number of subjects with a suspected diagnosis and the number of subjects in whom the diagnosis was not suspected

CONTACTS AND LOCATIONS:
Overall Officials: Federico Baronio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona:, Verona, Verona